CLINICAL TRIAL: NCT04609813
Title: Esophageal cAncer Screening Trial (EAST) Based on Novel Sponge Cytology：a Multicenter Nationwide Study
Brief Title: Esophageal cAncer Screening Trial
Acronym: EAST
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Collaborators: Shanghai Municipal Science and Technology Commission (Other Government)
Responsible Party: Principal Investigator, Zhaoshen Li, Director of Gastroenterology, Changhai Hospital
Other Study IDs: EAST
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Esophageal Squamous Cell Carcinoma; Esophageal Cancer; Gastroesophageal Junction Adenocarcinoma
Keywords: Esophageal Cancer; Screening and Early Detection; Sponge Cytology; Risk Stratification
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 1. Esophageal cell specimen collected with novel sponge cell collection device;
  2. Esophageal formalin-fixed paraffin-embedding tissue sample collected with endoscopic biopsy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Screening population: Participants underwent opportunistic endoscopic screening for esophageal cancer in high-risk regions in China will be enrolled in this study. Esophageal cell specimen will be collected by esophageal sponge cell collection device (Esoheal 1.0) prior to endoscopic examinations.
  Interventions: Diagnostic Test: Sponge cytological test

INTERVENTIONS:
Diagnostic Test: Sponge cytological test — Esophageal cell specimen were collected with Esoheal 1.0 sponge collection device. A prediction model will be built based on digital cytopathological features of participants.

SUMMARY:
This multicenter study aims to include 15000 participants undergoing screening upper gastrointestinal endoscopy and establish a risk prediction model for esophageal squamous cell carcinoma and esophagogastric junctional (EGJ) adenocarcinoma in high-risk areas. The prediction model will be built based on epidemiological and cytological features, acquired from the esophageal sponge cytology test. The primary study outcome is the diagnostic performance of the model to detect high-grade lesions (including carcinoma and high-grade intraepithelial neoplasia) of the esophagus and EGJ. Secondary outcomes include the number needed to screen, and dignostic performance of cytologist under AI assistance and abnornal cell count.

DETAILED DESCRIPTION:
Esophageal cancer is the seventh most common cancer and the sixth leading cause of cancer related death worldwide in 2020. The highest-incidence areas include Eastern and Central Asia, sub-Saharan Africa, and some South American countries, with esophageal squamous cell carcinoma (ESCC) being the dominant histologic subtype (nearly 90%). While esophageal adenocarcinoma, as a type of adenocarcinoma of the esophagogastric junction (AEG), was less common in these high-risk areas, but accounts for approximately two-thirds of esophageal cancer cases in Europe and North America. However, cardiac gastric cancer, another type of AEG, often shows high incidence in ESCC high-risk areas. Strikingly, 57.5% of global ESCC cases and 60.8% of cardiac gastric cancer cases were estimated to occur in China in 2018. Most esophageal cancer high-risk areas locate in developing countries with limited medical resources, high incidence and co-occurrence ESCC and AEG have posed significant challenges for disease control.

Both ESCC and AEG demonstrate dismal prognosis, with an overall 5-year survival of less than 30%. This is largely due to the asymptomatic nature of early-stage lesions, which frequently leads to delayed diagnosis. Population-based studies in China have confirmed that upper gastrointestinal endoscopy with Lugol's staining could increase the early detection rate and decrease both the incidence and mortality of ESCC and the mortality of AEG in very high-risk areas. However, the invasiveness and resource intensiveness of endoscopic procedure and relative low prevalence of target lesions in the general screening population (0.8% to 1.6%) limit its feasibility and cost-effectiveness in massive screening. Therefore, developing less invasive, readily accessible methods with acceptable diagnostic accuracy is urgently needed for enrichment of high-risk individuals prior to endoscopy. To date, few non-endoscopic preliminary screening methods were available for ESCC and AEG.

The esophageal sponge cytology is an emerging, minimally invasive, and convenient test for esophageal cancer as well as its precancerous lesions and conditions. The expandable sponge could harvest epithelial cells from the entire esophagus and the esophagogastric junction (EGJ) during withdrawn, and subsequent morphological or biomarker analysis could be performed. For Barrett esophagus (BE), the Cytosponge-trefoil factor 3 is a well-established non-endoscopic test, and could increase the detection of BE for 10.6-fold among patients with reflux symptoms in the primary care setting. For high-risk areas, where ESCC is the dominant subtype, several types of sponge cytology tests also gained promising yet preliminary results.

In our previous study, we have developed an artificial intelligence (AI)-assisted sponge cytology test, which automatically indicated potentially abnormal cells for cytologist diagnosis, and found the sensitivity and specificity to be 90.0% and 93.7% in community-based ESCC screening in China. However, the inadequacy of experienced cytologists makes this method still suboptimal for population-based screening, especially for resource-limited areas. Furthermore, AEG, which is also within the detection range of the sponge cytology, has not been investigated in previous studies. Therefore, we conducted the Esophageal cAncer Screening Trial (EAST) to develop and validate a fully-automated machine learning model based on cytological and epidemiological features for ESCC and AEG screening in high-risk areas.

ELIGIBILITY:
Inclusion Criteria:

* subjects underwent opportunistic endoscopic screening for esophageal cancer;
* aged 40-75 years.

Exclusion Criteria:

* subjects with alarming symptoms including dysphagia, hematemesis, and melena;
* subjects underwent upper endoscopy within 1 year;
* subjects with history of esophageal neoplasia;
* subjects with esophageal-gastric varices or esophageal stenosis;
* subjects with histories of esophageal or gastric surgery;
* subjects with coagulation disorders or taking anticoagulant or antiplatelet agents;
* subjects with other contraindications for upper endoscopy or biopsy;
* subjects with other serious disease or malignant tumor, and the life expectancy is less than 5 years;
* subjects that refuse to cooperate with data collection or sign the informed consent.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study enrolled participants undergoing endoscopic opportunistic screening for esophageal cancer, after excluding participants with alarming symptoms, known history of esophageal neoplasia, previous upper endoscopy within one year, and conditions that are not suitable for endoscopy and biopsy.
Sampling Method: Probability Sample
Enrollment: 14597 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance of the sponge cytology-based machine learning model for the main target lesions | through study completion, an average of 1.5 year
  The main target lesions include high-grade intraepithelial neoplasia and carcinoma of the esophagus and gastroesophageal junction.
  Diagnostic performance include AUC, average precision, sensitivity, specificity, positive predictive value, and negative predictive value.

SECONDARY OUTCOMES:
Diagnostic performance of cytologist under AI assistance | through study completion, an average of 1.5 year
  The main target lesions include high-grade intraepithelial neoplasia and carcinoma of the esophagus and gastroesophageal junction.
  Diagnostic performance include AUC, average precision, sensitivity, specificity, positive predictive value, and negative predictive value.
Numbers needed to screen | through study completion, an average of 1.5 year
  Numbers of participants needed to screen to prevent one main target lesion.
Diagnostic performance of abnormal cell count | through study completion, an average of 1.5 year
  The main target lesions include high-grade intraepithelial neoplasia and carcinoma of the esophagus and gastroesophageal junction.
  Diagnostic performance include AUC and average precision.

CONTACTS AND LOCATIONS:
Overall Officials: Zhao-Shen Li, MD, Study Director — Changhai Hospital; Luo-Wei Wang, MD, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
The IPD will not be made available to the public, but could be provided by the investigator on reasonable request.

REFERENCES:
- [Background] Gao Y, Xin L, Feng YD, Yao B, Lin H, Sun C, An W, Li ZS, Shi RH, Wang LW. Feasibility and Accuracy of Artificial Intelligence-Assisted Sponge Cytology for Community-Based Esophageal Squamous Cell Carcinoma Screening in China. Am J Gastroenterol. 2021 Nov 1;116(11):2207-2215. doi: 10.14309/ajg.0000000000001499. PMID 34546186
- [Derived] Bian Y, Xu Y, Chu C, Gao Y, Jiang H, Meng Q, Yu C, Zhou J, Li Z, Wang W, Lin H, Wang L. Accurate Nonendoscopic Detection of Early Esophageal Squamous Malignant Lesions Using Sponge-Based Methylated DNA Biomarkers. Am J Gastroenterol. 2025 Aug 22. doi: 10.14309/ajg.0000000000003745. Online ahead of print. PMID 40844617
- [Derived] Huang S, Gu X, Zhou H, Feng Y, Shi R, Wang W, Zhou A, Lin J. Application of Esophageal Sponge Cytology in Screening Esophageal Squamous Cell Carcinoma in a High-Risk Region of China. Cancer Med. 2025 Feb;14(3):e70467. doi: 10.1002/cam4.70467. PMID 39856802